CLINICAL TRIAL: NCT04132362
Title: Generating and Using Personalised Music Playlists to Improve Behavioural and Psychological Symptoms in People With Dementia: a Feasibility Study
Brief Title: Benefits of Personalised Music in Dementia - a Feasibility Study
Status: Recruiting | Type: Observational
Sponsor: Music for my Mind (Other)
Responsible Party: Sponsor
Other Study IDs: MFMM265263
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Dementia
Keywords: music; dementia; emotional responses
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People living with dementia, their families and carers: The cohort consists of people living with dementia. Each of them will be accompanied, throughout the study, by a family member or friend. They will take part together in a one hour music listening session, to discover their personalised playlist. Where possible, a care home staff member will join in, in order to witness the benefits of the music to the dementia resident and learn how to provide the music, as part of their care in the care home.
  Interventions: Behavioral: Personalised music listening; Behavioral: Using fMRI to investigate the effect of listening to personalised music evoking positive emotional response on brain activation; Behavioral: Personalised music listening in the community

INTERVENTIONS:
Behavioral: Personalised music listening — People will be sequentially recruited to discover their favourite music playlist, monitor their emotional responses to specific songs and explore the impact of listening to the music, on their behavioural and psychological symptoms. This will be done through a one hour music listening session, to discover the top 10-20 songs they respond to. It will then be followed by multiple shorter music listening sessions, initiated by the dementia resident themselves or their carer, where they listen to their favourite songs during their day, before difficult moments of care or during visits with their families.
Behavioral: Using fMRI to investigate the effect of listening to personalised music evoking positive emotional response on brain activation — 12 of the recruited participants, who have symptoms and signs of mild to moderate dementia will be invited to take part in this sub-study. Using an amended version of a previously employed fMRI paradigm, each study participant will be presented inside the MRI scanner with short 30 second epochs of music (identified as evoking a positive or neutral emotional response) in a block design. Each 30 second epoch of music will be followed by a 16 second period when participants will be asked to rate subjective changes in their affective state using a computerised visual analogue scale. Epochs of positive emotional stimuli will alternate with epochs of neutral emotional stimuli in a counterbalanced order of presentation in 2 runs of 10 epochs each (5 positive and 5 neutral in each run).
Behavioral: Personalised music listening in the community — 1000 families affected by dementia will be invited to use our WebApp to create a personalised playlist for their loved one with dementia and share their perceptions of how the music has affected the well-being of their loved one.

SUMMARY:
There is growing evidence for the benefits of music for individuals living with dementia but there has been limited research looking specifically at personalised music. Methodologies have not yet been developed to generate and play personalised music playlists quickly and cost effectively. The research team proposes a feasibility study to develop effective methodologies for:

i. efficient creation and delivery of personalised playlists for people with mild to moderate dementia in care homes; and

ii. assessing their responses to this music.

A long-list of personalised music (about 100 tracks) will be created by asking residents and their carers about the resident's musical tastes and background (particularly from their teenage years). A refined personalised playlist (of 10-20 tracks) will be created by playing excerpts from these tracks to the resident and gauging their responses including through direct feedback from the resident and their carer(s) plus observations of changes in facial expression, together with directly observed movements of hands, feet and/ or head, and changes in pulse rate (a monitor worn on the wrist to measure movement and pulse and the investigators will ask to film sessions). Care home staff and informal carers will use these playlists within the residents' care and the research team will use feedback from residents and carers to assess responses and explore whether factors such as the timing of listening or delivery methodology appear to affect the resident's well-being over time.

The findings from this study will be used to develop automated approaches to playlist creation (e.g. an App) and to inform further feasibility studies to: test and refine methodologies for use with participants with more advanced dementia; and explore more systematically the benefits of personalised music and factors that affect this, ultimately to inform the design of a subsequent larger scale intervention study.

Two substantial amendments were approved to this existing feasibility study on October 23, 2020. The two substantial amendments are:

1. To extend the main study to include participants who may lack capacity to consent.
2. A sub-study using fMRI to explore the mechanisms underlying reported beneficial effects of personalised music listening on behavioural and psychological symptoms in people living with dementia.

A further amendment was approved in January 2021, to recruit 1000 families affected by dementia, living at home or in the community, to use our recently developed WebApp to create a personalised playlist for their loved one living with dementia and provide their perceptions of how the music has impacted the well-being of the person with dementia.

DETAILED DESCRIPTION:
This research will adopt a mixed methods design for the study involving both quantitative and qualitative data collected and analysed simultaneously, then compared or related and interpreted.

Up to 10 participating care homes will be selected by Quantum Care Home Group in line with the inclusion/exclusion criteria. A total of 80 participating residents living with dementia, 80 informal carers and 20 care home staff will be selected from the participating care homes.

This study will explore:

1. The most effective and efficient methods for creating personalised playlists, including developing automated approaches, using technology (e.g. Apps and music recommendation algorithms).
2. The most easy-to-implement delivery methods for delivering personalised music to residents in care homes.
3. The most effective ways to assess responses to personalised music from people with dementia, including trialling automated analysis of changes in facial expression in video footage.
4. Initial impressions of whether factors such as timing of listening affect the observed impacts of listening to personalised music or whether listening prior to difficult care events appears to be beneficial (e.g. dressing, washing, toileting, sundowning, etc.).

A personalised playlist of about 100 songs will be created using responses to the music preferences questionnaire provided by the resident and their informal carer/Consultee/attorney (or paid carer). These questionnaires will be provided by the research team to the potential participants, identified by care home staff, together with the information pack and consent forms.

A music listening session will be arranged where the resident and their informal carer/Consultee/attorney will be played 30 seconds excerpts of each of the tracks (in 15 minute blocks over a period of up to 1 hour). The resident will be asked to wear a monitor on their wrist, similar to a watch, in order to monitor movement and pulse rate. The session will be filmed to enable analysis of emotional responses to music using machine learning analysis of changes in facial expression, as well as directly observed movements of hands, feet and/ or head. Where necessary the music listening session can be split into multiple shorter sessions to accommodate resident or care home requirements. Responses to the 30 second excerpts will be used to generate a refined personalised playlist for each participant, anticipated to be between 10 and 20 tracks.

The refined personalised playlists will be played to residents in music listening sessions throughout the duration of the study. How long music is played for and how frequently will, for the feasibility study, be determined by the resident, care home staff and/or informal carers. Different delivery methods for delivering personalised music will be tested including use of wireless headphones, smart speakers or other wireless speakers and their effectiveness and ease of use assessed through feedback from residents and focus groups and interviews with informal carers and care home staff. Duration and frequency of music listening sessions will, where possible, be logged through the listening history in the music app used and/or through data recorded by care home staff or informal carers.

A short training session will be provided in each participating care home to train staff and informal carers on delivering personalised music listening and collecting observational data (e.g. on timing of listening and observed effects on mood and behaviour). Fidelity, acceptability and appropriateness of the interventions will be assessed by the research team through the observation of selected personalised music listening sessions.

Approaches to assessing responses to the music that will be used include analysis of facial expression changes and movement in video footage, heart rate changes and qualitative information provided in reports from a member of the research team, residents, care home staff and/or informal carers. Impacts on well-being of residents over time will be assessed using scores derived from inventories for behavioural and psychological symptom assessment as a proxy, e.g. The Neuropsychiatric Inventory Nursing Home Version (NPI-NH), including for depression/apathy and anxiety/agitation. The Health-Related Quality of Life Measure for people living with dementia (DEMQOL) and DEMQOL-Proxy (administered with the informal carer/Consultee) will also be completed. It is expected that these tools will be used before the intervention and between 1 and 3 further times for each resident participant at appropriate intervals during the period of the study.

For this study the use of qualitative and quantitative assessment tools is for the purpose of developing and testing the appropriateness of personalised music listening and assessment methodologies rather than to draw conclusions about efficacy or otherwise of the intervention itself (which would be the subject of further studies subject to subsequent ethical approval). The quantitative data generated, therefore will only be used to supplement qualitative assessments to help infer/indicate factors for further investigation in subsequent feasibility studies and a longer-term larger scale intervention study i.e. to inform the design of those studies. Therefore, in this feasibility study, analysis of the quantitative measures is not intended to produce statistically significant data (the statistics involved will be mostly descriptive and, in some cases, inferential). Together with subsequent feasibility studies, it is intended to inform the design of the larger scale intervention study in which the sample size will be calculated to produce statistically significant results.

The study will trial the use of facial expression change through automated analysis of video footage. The initial pilot showed a strong correlation between the scores, indicating that, after further calibration, absolute thresholds can be derived to classify a track as either high or low response. Deep-learning facial expression change analysis will be developed to determine the feasibility or otherwise of using automated analysis of facial expression change in video footage. This will involve:

* Acquiring videos at 30 frames per second while music is played, extracting 1 image per second and generating 3 features for each.
* Performing face detection using Microsoft Azure Cognitive Services Application Programming Interface (API) and extracting an emotion score from the facial expression in 8 categories: anger, contempt, disgust, fear, happiness, neutral, sadness, and surprise. The research team will then form a secondary score based on a linear combination of these expressions and assign it to each frame.
* The research team will then aggregate the values of all frames acquired while a track was played to form a total response score by assigning different weights to the frames and deriving first-order statistics from the resulting distribution. The researchers can then compare the scores to subjective observation.

The views of care home staff and informal carers/Consultees/attorneys about the intervention will be sought throughout the study, via the means of focus group discussions and interviews. These focus group discussions and interviews will be conducted with care home staff and families in order to explore their views of how personalised playlists have an impact on residents including their impressions of the effect of variables such as timing of listening or the impact on difficult care situations. Direct feedback will also be sought from participating residents themselves, where feasible.

Informed consent for participation will be obtained, including for participation by informal carers/Consultees and care home staff, as well as residents. If anyone participating in the study, in any way indicates that they do not want to take part or in any way indicates that they are unhappy or distressed, then their participation will be paused (e.g. a different track played or a different question asked) and if the distress persists, the session will be stopped.

Informal carers/Consultees/attorneys will provide qualitative assessments of any benefits or disbenefits to them arising from the impact of personalised music listening on the behavioural and psychological symptoms of their relative/friend (e.g. improving relationship with carers and family). These assessments will be provided through participation in structured focus groups. Informal carers/Consultees/attorneys will participate in up to 3 focus groups, conducted by a member of the research team, experienced in qualitative research, once the refined personalised playlist is completed, between 2 and 4 months later and at the conclusion of their participation in the study.

Care home staff will provide qualitative assessments of any benefits or disbenefits to them arising from the impact of personalised music listening on the behavioural and psychological symptoms of the resident, for example:

* improving relationship with carers and family;
* improved quality or ease of care provision such as easing of distress caused by difficult care events.; and
* ease of incorporation of personalised music therapy into the usual working practices of the care homes.

These assessments will be provided through participation in structured focus groups. Care home staff will participate in up to 3 focus groups, conducted by a member of the research team, experienced in qualitative research, once the refined personalised playlist is completed, 2-4 months afterwards and at the conclusion of their participation in the study. If the care home staff are unable to participate in a focus group, a semi-structured 1:1 interview will be conducted instead.

As individuals with more severe dementia may lack the capacity to communicate their music preference or emotional responses to listening to music, this study will both:

* explore using the outcome measures as an objective way of gauging their preferences and responses by comparing responses measured through biomarkers and subjective assessments given by individuals living with less severe stages of dementia and their carers, family and/or friends; and
* work directly with people with advanced dementia who are not able to communicate their music preferences or emotional responses to listening to music, instead gathering such information from their carers, family and/or friends and measuring responses through biomarkers and subjective assessments given by these individuals.

The eventual larger scale study will explore issues of cost effectiveness, in addition to clinical effectiveness.

Pilot sub-study: Benefits of personalised music in dementia - a pilot study to investigate mechanisms of action

12 of the 80 participants (who have capacity to provide informed consent) will be further invited to take part in a pilot sub-study to investigate mechanisms of action.The capacity of residents to give consent will be assessed and documented by care home staff. The participants will be provided with an information sheet about the sub-study, consent forms and an MRI Safety Screen Questionnaire. This pilot study will help develop the mechanistic rationale for a larger scale intervention study to explore the effects of personalised music on behavioural and psychological symptoms in people with dementia.

In January 2021 we received approval to add a sub-study to this project, to use a Music for my Mind developed Web Application (the App), to invite relatives, friends or carers of a person living with dementia to use the App to create and deliver a personalised music playlist to their loved one and seek their feedback on the use of the technology and how it can be improved, and on their perceptions of how listening to the playlist has impacted on the well-being of the person living with dementia and, by extension, their own well-being.

This App has been developed as a lateral response to the Covid-19 epidemic (since the main study cannot currently be progressed, as it requires access to care homes). Our overall goal is to benefit people living with dementia and this sub-study aims to explore new ways of achieving that.

The participants in this sub-study will be the relatives, friends and/or carers of people living with dementia (whether the person living with dementia lives in a care home, their own home or with a relative). The planned sample size is 1000 participants. The participants will be recruited entirely through digital means through our team and supporter networks; through local radio and local branches of partner charities; through social media.

ELIGIBILITY:
Inclusion Criteria:

A care home meeting all of the following criteria will be eligible to join the feasibility studies:

* Is located in South East England;
* Has at least 5 residents who care home staff estimate to be eligible for the studies;
* Agrees to identify a suitable space for personalised music listening to be trialled;
* Agrees to make staff available to select residents and support the studies;

A resident meeting all of the following criteria will be eligible to participate in the feasibility studies:

* A permanent resident within a care home run by the Quantum Care Home Group;
* Has been assessed by suitably qualified/trained care home staff (or a medical professional) as having symptoms and signs of dementia (of any type).
* Has one or more family member/carer willing to participate in this study by providing sufficient responses to a questionnaire about the resident's musical preferences and background and feedback on the resident's responses to listening to personalised music.
* Has the ability to communicate in English; and
* For participants who are assessed as lacking mental capacity to consent to participation, has an attorney or Consultee willing to support their inclusion in the study.

An informal carer meeting all of the following criteria will be eligible to participate in the feasibility studies:

* People above the age of 18 who are a family member or friend and act as an informal carer for a participant with dementia.
* Has the ability to communicate in English.

A care home staff meeting the following criteria will be eligible to participate in the feasibility study:

* Health and social care staff, paid to provide care to individuals with dementia within participating care homes. This may include Managers, Registered Nursing staff, Care Assistants or Activity Coordinators.
* Has the ability to communicate in English.

Exclusion Criteria:

A care home meeting any of the following criteria will not be eligible to join the feasibility study if it is:

* Rated at the last Care Quality Commission (CQC) inspection as Needs Improvement or Inadequate;
* Subject to CQC enforcement notices, admission bans or major CQC compliance issues;
* Currently, or has recently been involved in, another research study or trial that conflicts with personalised music or with data collection during the course of these studies.

A resident meeting any of the following criteria will not be eligible to participate in the feasibility studies:

* Assessed by care home staff or a medical professional as having severe depression;
* Assessed as being unable to hear music through headphones;
* Is so severely physically impaired as to make it unlikely that the researchers, carers or informal carers will be able to observe responses to personalised music through (for example, changes in facial expression, tapping of feet or fingers etc)
* Is currently, or has recently been involved in, another research study or trial that conflicts with personalised music listening or with data collection during the course of these studies;
* Is expected to die before the completion of their participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 80 residents living with dementia, from up to 10 different care homes. Up to 80 informal carers, participating in music listening sessions, focus groups and/or providing feedback.
  Up to 20 care home staff, participating in focus groups or interviews. In addition, all staff in participating care homes will participate in administration of personalised music interventions.
  Up to 1000 families affected by dementia living at home or in the community.
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Median time (in hours) required to generate personalised music playlists for participants living with dementia assessed using activity logs recorded by researchers, carers and/or relatives/friends. | 6 months per participant
  The primary outcome sought is the ability to generate a personalised playlist for a person living with dementia requiring an aggregate time input from the researchers, relatives/friends and/or their paid carer(s) of under 2 hours. This time input will consist of the time required to complete the music preferences questionnaire and the total elapsed time of the music listening session. During that music listening session, excerpts of tracks from a long list of 100 songs generated form the questionnaire responses are played to the person living with dementia and those tracks that elicit the strongest positive responses will be included in their final personalised playlist. The time required for each of these tasks will be recorded in activity logs by the researchers, carers and/or relatives/friends of the person living with dementia.
Acceptability by participants of the delivery method(s) of personalised playlists in care homes, assessed through qualitative methods such as feedback from participants (people living with dementia, their relatives/friends and their carers). | 6 months per participant
  A range of different methods will be tested to deliver (play) personalised music playlists once they are generated. The acceptance (or otherwise) of these methods (e.g. use of headphones, smart speakers, etc) will be assessed through qualitative research by gathering feedback from participants (people living with dementia, their relatives/friends and their carers) including from activity logs completed by carers and/or relative/friends, focus groups with carers and relative/friends and interviews with participants.

SECONDARY OUTCOMES:
Extent of correlation between measures of emotional responses of people living with dementia to personalised music listening (using facial expression change algorithm) with direct observation by researchers, documented in activity logs. | 6 months per participant
  The effectiveness (or otherwise) of machine learning analyses of changes in facial expression (using Microsoft Azure Cognitive Services Application Programming Interface with video recordings of music listening sessions) to derive quantitative measures of emotional responses to music listening will be assessed through analysis of the extent of correlation of these machine learning derived measures with direct observations of responses by researchers. Such observations will be recorded manually during the music listening session at which excerpts of the long list of tracks is played and will include observations of changes in pulse rate (measured with an Empatica 4 device) and of responses such as singing, dancing, smiling and movement of hands, feet or head.
Assessing the feasibility of acquiring functional magnetic resonance imaging (fMRI) data while listening to personalised music | 4 months per participant
  Through the pilot sub-study, to explore the feasibility of acquiring functional magnetic resonance imaging (fMRI) data while listening to personalised music to obtain:
  * evidence to contribute to hypothesis generation that listening to personalised music evocative of a positive emotional state engages brain regions implicated in BPSD and that the effect on brain activation in key regions of interest (ROI) is in a direction that is consistent with a potential beneficial effect on BPSD; and
  * estimates of effect-size that may inform a future larger scale intervention study.

OTHER OUTCOMES:
Number of participants who exhibit improved well-being following a period of listening to personalised playlists as part of their care package, measured through changes in quality of life measures and Behavioural and Psychological Symptoms as a proxy. | 6 months per participant
  Reductions (or otherwise) in Behavioural and Psychological Symptoms (anxiety/agitation, depression/apathy, etc) will be assessed using qualitative research methods to analyse feedback from participants (people living with dementia, their relatives/friends and their carers) including from activity logs completed by carers and/or relatives/friends, focus groups and/or interviews with carers, participants and their relatives/friends. These measures will be combined with quantitative ones including responses to the Neuropsychiatric Inventory Questionnaire and biomarkers such as changes in facial expression, pulse rate. Analyses of these data will be used to indicate whether variables such as the timing of listening to personalised music (how frequently, what time of day and whether it is before, during or after a difficult care event) affect the extent to which participants' well-being improves (or otherwise), using assessment of Behavioural and Psychological Symptoms as a proxy.

CONTACTS AND LOCATIONS:
Overall Officials: Keith McAdam, Principal Investigator — Music for my Mind
Locations (1):
- Willow Court, Harpenden, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No